CLINICAL TRIAL: NCT02883959
Title: Evaluation of the Analgesic Effect of Music Therapy in Critically Ill Patients During Potentially Painful Nursing Procedures: a Pilot Study
Acronym: Painkiller
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, LEGRIEL stephane, Study principal investigator, Versailles Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12/18_Painkiller
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Pain
Keywords: critically ill; mechanical ventilation; pain; nursing; music
MeSH Terms: conditions — Pain; Critical Illness | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- music therapy (Experimental): Music therapy
  Interventions: Other: music therapy
- control arm (No Intervention): No music

INTERVENTIONS:
Other: music therapy — Music therapy will be delivered through headphones during nursing procedures (toilet and/or surgical dressings): from initiation up to 30 minutes after the end of procedure.
  Arms: music therapy

SUMMARY:
Pain is a common problem encountered in about 60 % of critically ill patients who can communicate. Its occurrence can be related to several causes, mainly dominated by invasive procedures.

Pain management is typically based on a combination of prevention, evaluation, and therapeutic agents. However, it appears important to develop adjuvant approaches. Music therapy is one of them and that has been evaluated in various medical conditions.

The aim of our study is to evaluate the analgesic effect of music therapy in critically ill patients during potentially painful nursing procedures.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age≥18 years) hospitalized in Intensive Care Unit
* Requiring mechanical ventilation
* Who cannot communicate
* With a Richmond Agitation Sedation Scale (RASS) score [-3; +4]

Exclusion Criteria:

* Age < 18 years
* Receiving neuromuscular blockade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
proportion of pain exposure during nursing procedures | 150 minutes
  total length of pain exposure to a BPS score over or equal to 5 divided by total length of nursing procedure

SECONDARY OUTCOMES:
proportion of maximal pain exposure during nursing procedures | 150 minutes
  Total length of exposure to the maximal BPS score (over or equal to 5) among total length of nursing procedure

CONTACTS AND LOCATIONS:
Locations (1):
- CH Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacq G, Melot K, Bezou M, Foucault L, Courau-Courtois J, Cavelot S, Lang A, Bedos JP, Le-Boeuf D, Boussard JM, Legriel S. Music for pain relief during bed bathing of mechanically ventilated patients: A pilot study. PLoS One. 2018 Nov 14;13(11):e0207174. doi: 10.1371/journal.pone.0207174. eCollection 2018. PMID 30427906